CLINICAL TRIAL: NCT06854120
Title: Body Surface Gastric Mapping in Patients With Dyspeptic Symptoms: Recordings at Baseline and on Medical Therapy
Brief Title: Prokinetics and Body Surface Gastric Mapping in Dyspeptic Patients: Baseline and Treatment Effects
Status: Not yet recruiting | Type: Observational
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: University of Western Sydney (Other); Temple University (Other); North Shore Hospital, New Zealand (Other)
Responsible Party: Principal Investigator, Greg O'Grady, MD/PhD, University of Auckland, New Zealand
Other Study IDs: AK-PRO-001
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gastroparesis; Functional Dyspepsia
Keywords: Gastroparesis; Functional Dyspepsia; Gastric Motility; Body Surface Gastric Mapping
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment: Patients undergoing Body Surface Gastric Mapping before and after administration of prescribed prokinetic/neuromodulator
  Interventions: Device: Gastric Alimetry

INTERVENTIONS:
Device: Gastric Alimetry — The Gastric Alimetry™ System is intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of various gastric disorders.

SUMMARY:
Functional dyspepsia and gastroparesis are common stomach disorders with symptoms like early satiety, nausea, and abdominal pain, and are often evaluated with gastric emptying tests, although the correlation with symptoms is weak. Prokinetic agents (e.g., metoclopramide, erythromycin) and symptom modulators (e.g., nortriptyline, mirtazapine) are commonly used, but selecting the right medication can be difficult, as it's often based on symptoms rather than the underlying gastric issues. Body Surface Gastric Mapping (BSGM) using the Gastric Alimetry device is a novel, non-invasive tool to assess gastric myoelectrical activity and symptoms. This study aims to perform two BSGM recordings-one before and one after medical therapy-to understand how medications affect gastric function and identify baseline BSGM factors that could predict responses to treatment, potentially guiding tailored therapies based on individual gastric dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Diagnosis of gastroparesis and/or functional dyspepsia
* Being prescribed a prokinetic agent or symptom modulator for their clinical care
* Able to undergo BSGM recording both before and during treatment
* Able to give informed consent for undergoing a baseline BSGM recording and an additional recording while on treatment

Exclusion Criteria:

* Under 18 years of age
* Prior surgery on esophagus, stomach (appendectomy and cholecystectomy are allowed)
* History of skin allergies or a history of extreme sensitivity to cosmetics or lotions
* Pregnant women
* No vulnerable groups such as prisoners, individuals with known cognitive impairment, or institutionalized individuals be involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastroparesis and/or functional dyspepsia who are prescribed prokinetics/neuromodulators.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-02-26 (Estimated); Primary Completion 2028-02-26 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Change in overall postprandial BSGM Gastric Alimetry Rhythm Index (minimum: 0; maximum: 1) on treatment compared to baseline (with a lower score meaning worse outcome). | 8 weeks

SECONDARY OUTCOMES:
Change in overall BSGM BMI-Adjusted Amplitude on treatment compared to baseline (normal range: 22-70 μV). | 8 weeks
Change in overall BSGM Principal Gastric Frequency (minimum: 0; maximum: 5) on treatment compared to baseline (normal range: 2.65-3.35 cpm). | 8 weeks
Change in overall BSGM Fed:Fasted Amplitude Ratio on treatment compared to baseline (normal range: >1.08). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Principal Investigator — Temple University; Vincent Ho, MBBS, FRACP, FACP, PhD, Principal Investigator — University of Western Sydney; Charlotte Daker, MD, Principal Investigator — University of Auckland, New Zealand; Greg O'Grady, MD, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (3):
- Temple University, Philadelphia, Pennsylvania, United States
- Western Sydney University, Sydney, New South Wales, Australia
- Te Whatu Ora Waitemata, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
The study design means that no identifiable data will be shared beyond immediate study researchers at each location.

REFERENCES:
- [Background] Varghese C, Schamberg G, Calder S, Waite S, Carson D, Foong D, Wang WJ, Ho V, Woodhead J, Daker C, Xu W, Du P, Abell TL, Parkman HP, Tack J, Andrews CN, O'Grady G, Gharibans AA. Normative Values for Body Surface Gastric Mapping Evaluations of Gastric Motility Using Gastric Alimetry: Spectral Analysis. Am J Gastroenterol. 2023 Jun 1;118(6):1047-1057. doi: 10.14309/ajg.0000000000002077. Epub 2022 Dec 20. PMID 36534985
- [Background] Wang WJ, Foong D, Calder S, Schamberg G, Varghese C, Tack J, Xu W, Daker C, Carson D, Waite S, Hayes T, Du P, Abell TL, Parkman HP, Huang IH, Fernandes V, Andrews CN, Gharibans AA, Ho V, O'Grady G. Gastric Alimetry Expands Patient Phenotyping in Gastroduodenal Disorders Compared with Gastric Emptying Scintigraphy. Am J Gastroenterol. 2024 Feb 1;119(2):331-341. doi: 10.14309/ajg.0000000000002528. Epub 2023 Oct 30. PMID 37782524
- [Background] Gharibans AA, Calder S, Varghese C, Waite S, Schamberg G, Daker C, Du P, Alighaleh S, Carson D, Woodhead J, Farrugia G, Windsor JA, Andrews CN, O'Grady G. Gastric dysfunction in patients with chronic nausea and vomiting syndromes defined by a noninvasive gastric mapping device. Sci Transl Med. 2022 Sep 21;14(663):eabq3544. doi: 10.1126/scitranslmed.abq3544. Epub 2022 Sep 21. PMID 36130019